CLINICAL TRIAL: NCT00923949
Title: Pilot Trial of Pioglitazone in Adults Undergoing Surgical Resection of Non-Small Cell Lung Cancer
Brief Title: Pioglitazone to Treat Adults Undergoing Surgery for Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never published; terminated early due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Giuseppe Giaccone, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080208; 08-C-0208; NCT00751725 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2012-02

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC Stage Ia-IIb; Resectable NSCLC; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental): 45 mg tablet daily by mouth for six weeks
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 45 mg tablet daily by mouth for six weeks

SUMMARY:
Background:

* Pioglitazone is a drug that belongs to the class of antidiabetic agents called thiazolidinediones. It is approved for treatment of type 2 diabetes mellitus.
* Research suggests that the thiazolidinediones may have anticancer activity that can reduce cancer risk or cause tumors to shrink.

Objectives:

-To test how a pioglitazone works as a treatment of Stage IA to IIB Non-Small Cell Lung Cancer (NSCLC) and to look at the effect of the drug on cancer cells.

Eligibility:

-Patients 18 years of age or older who will undergo surgery for Stage IA to IIB non-small cell lung cancer (NSCLC).

Design:

-The study includes a screening visit to determine eligibility, treatment with pioglitazone, a follow-up visit after 2 to 3 weeks of treatment and a post-surgery visit. Procedures include:

1. Medical history, physical examination, blood tests, electrocardiogram
2. Bronchoscopy to obtain cancer cells. This is done before pioglitazone treatment begins and again during lung surgery. Some patients may also require mediastinoscopy or biopsy to collect cells.
3. Treatment with pioglitazone tablets once a day for at least 2 weeks and no more than 6 weeks, depending on when surgery has been scheduled.
4. Positron emission tomography (PET) scan before starting pioglitazone treatment. National Cancer Institute (NCI) patients also have a follow-up PET scan after treatment but before surgery.

DETAILED DESCRIPTION:
Background:

Lung cancer is the leading cause of cancer deaths in the United States (US). Chemoprevention is an active area of investigation for reducing the burden of this disease. However, the choice of chemopreventive targets requires sufficient human data to justify extensive clinical interventions.

Peroxisome proliferator-activated receptor gamma (PPAR gamma) is a ligand activated nuclear transcription factor that is a key regulator of adipogenic differentiation. PPAR gamma ligands, particularly the thiazolidinedione class of antidiabetic agents exemplified by pioglitazone, are under investigation as chemopreventive agents.

PPAR gamma is expressed in normal lung and in NSCLC. PPAR gamma ligands induce apoptosis in NSCLC cell lines and modulate their differentiation status. Animal carcinogenesis studies, however, show equivocal efficacy in prevention of lung cancer.

Relevant human data are limited to an epidemiologic study showing that lung cancer risk is decreased in diabetics taking thiazolidinediones and a small phase IIa trial of pioglitazone in oral leukoplakia showing an 80% clinical response (partial response (PR)+ complete response (CR)). Further data are needed prior to engaging in a phase II lung chemoprevention trial.

Objectives:

The objectives of this pilot feasibility study are to evaluate the effect of pioglitazone on the expression of multiple biomarkers in NSCLC tumor tissue and in histologically normal and premalignant tissue.

* The primary endpoint will be the effect of pioglitazone on Ki-67, a marker of proliferation, in tumor tissue.
* The secondary objectives are to determine the effects of pioglitazone on multiple biomarkers in tumor, premalignant, and histologically normal bronchial epithelium and in serum:

  * Tumor tissue biomarkers: apoptotic index (AI), cyclin D1, p21/Waf1, PPAR gamma, mucin 1 (MUC1), gelsolin, proline oxidase, 15-hydroxyprostaglandin dehydrogenase (15-PGDH)
  * Premalignant tissue biomarkers: Ki-67, apoptotic index, PPAR gamma
  * Histologically normal tissue biomarkers: Ki-67, PPAR gamma
  * Serum markers affected by pioglitazone; C-reactive protein, CA 15-3
  * Serum tumor markers: carcinoembryonic antigen (CEA), cancer antigen 125 (CA-125)
* Additional secondary objectives are:

  * To evaluate the toxicity and safety of pioglitazone in this patient population,
  * To determine if limited treatment with pioglitazone affects tumor metabolic activity as determined by fludeoxyglucose positron-emission tomography (FDG-PET).

Eligibility:

Adult patients with newly diagnosed histologically confirmed stage Ia-IIb resectable non-small cell lung cancer who are eligible for and scheduled to undergo definitive surgery.

Eastern Cooperative Oncology Group (ECOG) 0-2

Normal organ function

Design:

Open label, multi-center, non-randomized pilot study to evaluate the effect of pioglitazone on the expression of multiple biomarkers in NSCLC tumor tissue and in histologically normal and premalignant tissue obtained from treatment-naive individuals who will receive oral pioglitazone prior to definitive surgery. The primary endpoint is Ki-67 measured in tumor tissue.

Patients will receive pioglitazone 45 mg po qd for a minimum of 2 weeks or a maximum of 6 weeks, with duration of treatment determined by standard of care and scheduling of surgery.

The study will consist of a screening visit, baseline bronchoscopy with tissue acquisition, pioglitazone treatment for 2-6 weeks, a 2-week on-treatment clinic visit, definitive surgical resection with bronchoscopy performed at the time of resection, and a post-surgery visit. Tissue (visually normal and abnormal areas identified during bronchoscopy) and tumor will be obtained at baseline and at the time of surgery. Patients who receive their treatment at NCI will also undergo a follow up FDG-PET scan after a minimum of 2 weeks of pioglitazone treatment.

Up to 25 patients are expected to be enrolled to identify 20 patients with adequate tissue for biomarker analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult patients with newly diagnosed stage Ia-IIb resectable non-small cell lung cancer who will be undergoing definitive surgery. If histologic confirmation of lung cancer has not previously been made, the baseline study bronchoscopy, as outlined in section 3.6.2, or computed tomography (CT)-guided biopsy with tissue saved for protocol use may be used to document NSCLC, after obtaining informed consent. Should the bronchoscopy or CT-guided biopsy be negative for non-small cell lung cancer (NSCLC), the patient will be taken off study prior to drug treatment. At National Cancer Institute (NCI), histologic confirmation of the diagnosis will be performed by the NCI Laboratory of Pathology.
  2. Age greater than or equal to 18 years of age.
  3. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
  4. Patients must have the capacity and willingness to sign a written informed consent and demonstrate willingness to comply with an oral regimen.
  5. The time between initial diagnosis and the scheduled surgery date allow for the subject to receive a minimum of 2 weeks or a maximum of 6 weeks treatment with pioglitazone. The maximum time between enrollment on this trial and surgery will be 6-weeks and there will be no delay between the end of pioglitazone treatment and surgery.
  6. Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,500/mL
* hemoglobin greater than 10 g/dL
* platelets greater than or equal to 100,000/mL
* Bilirubin less than 1.8 mg/dL
* aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than 1.5 times upper limits of institutional normal
* creatinine less than 1.5 times upper limit of institutional normal

  7. Patients must agree to swallow oral tablets.

  8. Patients who will agree to undergo two bronchoscopies as detailed in section 3.6.2 (before treatment and at the time of surgery).
* For those patients who are undergoing mediastinoscopy as part of their standard-of-care, the pre-treatment bronchoscopy may be performed during the mediastinoscopy. If the patient remains eligible for definitive surgical resection after the mediastinoscopy, the patient may begin pioglitazone treatment on this protocol.

  9. Females are eligible to participate in the study if
* She is of non-childbearing potential as defined by having had a hysterectomy, a bilateral oophorectomy, a bilateral tubal ligation, or having been post-menopausal for greater than or equal to 1 year.
* She is of childbearing potential and has a negative pregnancy test within 2 weeks of the starting the study drug and agrees to the use of non-hormonal methods of birth control, e.g., barrier methods, for the duration of the study due to possible drug interactions.

EXCLUSION CRITERIA:

1. Pregnant or lactating women.
2. Patients who are undergoing chemotherapy, treatment with biologic agents, or radiation therapy. Prior chemotherapy, biologic agent treatment, or radiation therapy, greater than 1 year ago, is allowed.
3. Patients with greater than or equal to class II New York Heart Association (NYHA) congestive heart failure or history of congestive heart failure.
4. Patients with greater than or equal to grade 2 (moderate) edema.
5. Patients with diabetes mellitus being treated with insulin or any pharmacologic therapy.
6. Patients taking gemfibrozil or rifampin, due to drug interactions with pioglitazone.
7. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active liver disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - New York University, New York, New York

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Elstner E, Muller C, Koshizuka K, Williamson EA, Park D, Asou H, Shintaku P, Said JW, Heber D, Koeffler HP. Ligands for peroxisome proliferator-activated receptorgamma and retinoic acid receptor inhibit growth and induce apoptosis of human breast cancer cells in vitro and in BNX mice. Proc Natl Acad Sci U S A. 1998 Jul 21;95(15):8806-11. doi: 10.1073/pnas.95.15.8806. PMID 9671760
- [Background] Sarraf P, Mueller E, Jones D, King FJ, DeAngelo DJ, Partridge JB, Holden SA, Chen LB, Singer S, Fletcher C, Spiegelman BM. Differentiation and reversal of malignant changes in colon cancer through PPARgamma. Nat Med. 1998 Sep;4(9):1046-52. doi: 10.1038/2030. PMID 9734398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 participant was accrued to this study.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Ki-67 Due to the Effect of Pioglitazone in Tumor Tissue
Description: Antigen ki-67 (Ki-67) will be assessed by immunohistochemistry.
Time Frame: 58 days
Population: No participants were analyzed because only one participant went on study and he did not undergo the requisite lung cancer resection due to disease progression, which means there was insufficient tissue to perform all the secondary tumor marker analyses. There is no statistical power to draw any conclusions and thus the data are not informative.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Effects of Pioglitazone on Multiple Biomarkers in Tumor
Description: Apoptotic index (A1) will be assessed by terminal deoxynucleotidyl transferase dUTP end labeling (TUNEL) and cyclin D1, p21/Waf1, PPARy, MUC1, gelsolin, proline oxidase, and 15-hydroxyprostaglandin dehydrogenase (15-PGDH) will be assessed by immunohistochemistry.
Time Frame: 58 days
Population: as for outcome 1
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For details about the adverse events see the adverse event module.
Time Frame: 58 days
Measure: Number; unit: Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Number of Participants With Metabolic Activity Determined by Fludeoxyglucose Positron-emission Tomography (FDG-PET)
Description: Response will be evaluated by FDG-PET. Response is defined as a decrease of standardized uptake values (SUV) of more than one.
Time Frame: 58 days
Population: as for outcome 1
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Effects of Pioglitazone on Premalignant Tissue Biomarkers
Description: Premalignant tissue biomarkers ki-67, apoptotic index and peroxisome proliferator-activated receptor gamma (PPARgamma) will be assessed by immunohistochemistry.
Time Frame: 58 days
Population: as for outcome 1
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Effects of Pioglitazone on Histologically Normal Tissue Biomarkers
Description: ki-67 and peroxisome proliferator-activated receptor gamma (PPARgamma) will be assessed by immunohistochemistry.
Time Frame: 58 days
Population: as for outcome 1
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Effects of Pioglitazone on Serum Tumor Markers
Description: C-reactive protein, cancer antigen 15-3 (CA 15-3), cancer antigen 125 (CA-125) and carcinoembryonic antigen (CEA) will be assessed by immunohistochemistry.
Time Frame: 58 days
Population: as for outcome 1
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 58 days
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study never published; terminated early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No